CLINICAL TRIAL: NCT03247075
Title: Internet-delivered Cognitive Behavior Therapy Versus Internet-delivered Support and Counseling for Youth With Social Anxiety Disorder - A Randomized Controlled Trial
Brief Title: Internet-delivered CBT vs Internet-delivered Support and Counseling for Youth With Social Anxiety Disorder - An RCT
Acronym: SOFT RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Eva Serlachius, Associate professor, child psychiatrist, MD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DNR 2017/1027-31/2
Record Dates: First submitted 2017-08-08; First posted 2017-08-11 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Social Anxiety Disorder
Keywords: Social anxiety disorder; Cognitive Behavior Therapy; Internet-delivered treatments; Children and adolescents; Randomized controlled trial
MeSH Terms: conditions — Phobia, Social | interventions — Cognitive Behavioral Therapy; Palliative Care; Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-delivered Cognitive Behavior Therapy (Experimental): 10 weeks of guided Internet-delivered Cognitive Behavior Therapy
  Interventions: Behavioral: Cognitive Behavior Therapy
- Internet-delivered Support and Counseling (Active Comparator): 10 weeks of guided Internet-delivered support and counseling
  Interventions: Behavioral: Support and Counseling

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy — Guided Internet-delivered CBT includes exposure training, coping techniques and cognitive components, intended to reduce social anxiety symptoms
  Arms: Internet-delivered Cognitive Behavior Therapy
Behavioral: Support and Counseling — Guided Internet-delivered support and counseling includes educative material about social anxiety and health related issues such as physical activity, nutritious diet, sleep habits etc.
  Arms: Internet-delivered Support and Counseling

SUMMARY:
Social anxiety disorder among youth is highly prevalent and causes significant impairment in the lives of the affected. In spite of cognitive behavior therapy (CBT) being an effective treatment, research suggests that many young people with this disorder do not have access to good-quality CBT. Internet-delivered CBT could be an effective method to increase availability of evidence-based treatments for youth with social anxiety disorder. The primary objective of this study is to test the efficacy of internet-delivered CBT (ICBT) for youth (10 - 17 years) with social anxiety disorder. The investigators aim to conduct a randomized controlled trial with N = 101 participants. Participants will be randomized to either the active treatment arm (guided ICBT) or to a control condition (guided internet-delivered support and counseling). Follow-ups will be conducted at 3 and 12 months after post-assessment.

ELIGIBILITY:
Inclusion Criteria:

* A principal diagnosis of social anxiety disorder, as defined by DSM-5
* Age between 10 and 17 years
* Ability to read and write Swedish
* Daily access to the internet through a computer or similar device
* A parent or caregiver that is able to co-participate in the treatment
* Participants on psychotropic medication must have been on a stable dose for the last 6 weeks prior to baseline assessment

Exclusion Criteria:

* Diagnosed with autism spectrum disorder, psychosis, bipolar disorder or severe eating disorder
* Present risk of suicide
* Ongoing alcohol or substance abuse
* Occurrence of domestic violence
* Completed CBT for any anxiety disorder within the last 6 months (defined as at least 5 sessions of CBT including in vivo exposure sessions)

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Clinician Severity Rating (CSR) | 6 months (14 months including follow-up)
  A 0-8 rating by a professional assessor, specifying the severity of social anxiety

SECONDARY OUTCOMES:
Anxiety Disorder Interview Schedule for DSM-IV, child and parent versions (ADIS C/P) - Social anxiety disorder | Measured over the course of 6 months (14 months including follow-up)
  Diagnostic status: Social anxiety disorder
Anxiety Disorder Interview Schedule for DSM-IV, child and parent versions (ADIS C/P) - Comorbid disorders | Measured over the course of 6 months (14 months including follow-up)
  Diagnostic status: Comorbid psychiatric disorders
Clinical Global Impression - Improvement (CGI-I) | Measured over the course of 3 months (12 months including follow-up)
  A 1-7 rating by a professional assessor, specifying the degree of improvement from treatment
Children's Global Assessment Scale (CGAS) | Measured over the course of 6 months (14 months including follow-up)
  A 0-100 rating by a professional assessor, specifying global functioning
Liebowitz social anxiety scale for children and adolescents (LSAS-CA) - Child version | 6 months (14 months including follow-up)
  A self-rated measure of severity of social anxiety
Liebowitz social anxiety scale for children and adolescents (LSAS-CA) - Parent version | Measured over the course of 6 months (14 months including follow-up)
  A parent-rated measure of severity of social anxiety
Revised Children´s Anxiety and Depression Scale - (RCADS) - Parent version | Measured over the course of 6 months (14 months including follow-up)
  A parent-rated measure of severity of anxiety and depression
Revised Children´s Anxiety and Depression Scale - (RCADS) Depression sub scale - Child version | Measured over the course of 6 months (14 months including follow-up)
  A parent-rated measure of severity of anxiety and depression
Anticipatory social behaviors scale (ASBQ) | Measured over the course of 6 months (14 months including follow-up)
  A self-rated measure of anticipatory anxiety before social situations
Post-event processing questionnaire revised (PEPQ-R) | Measured over the course of 6 months (14 months including follow-up)
  A self-rated measure of anxiety and rumination experienced after social situations
Focus of attention questionnaire (FAQ) | Measured over the course of 6 months (14 months including follow-up)
  A self-rated measure of self-focus in social situations
The Subtle Avoidance Frequency Examination (SAFE) | Measured over the course of 6 months (14 months including follow-up)
  A self-rated measure of safety behaviors in social situations
The Child Health Utility 9D (CHU 9D) - Child version | Measured over the course of 6 months (14 months including follow-up)
  A self-rated measure of quality of life
Client Satisfaction Questionnaire (CSQ-) - Child version | Measured only at post-treatment
  A self-rated measure of treatment satisfaction
Client Satisfaction Questionnaire (CSQ-) - Parent version | Measured only at post-treatment
  A parent-rated measure of treatment satisfaction
Treatment credibility and expectancy - Child version | Measured at one time-point, at week three in the allocated intervention.
  A self-rated measure of credibility and expectancy of allocated treatment condition
Treatment credibility and expectancy - Parent version | Measured at one time-point, at week three in the allocated intervention.
  A parent-rated measure of credibility and expectancy of allocated treatment condition
Education, Work and Social Adjustment Scale (EWSAS) - Parent version | Measured over the course of 6 months (14 months including follow-up)
  A parent-rated measure of functioning in everyday life
Hospital Anxiety and Depression Scale (HADS) | Measured only at pre-treatments
  A self-rated measure of anxiety and depression among parents
Alcohol Disorder Identification Test (AUDIT) | Measured over the course of 6 months (14 months including follow-up)
  A self-rated screening measure for hazardous and harmful alcohol consumption
Drug Use Disorders Identification Test (DUDIT) | Measured over the course of 6 months (14 months including follow-up)
  A self-rated screening measure for drug-related problems
Family Accommodation Scale-Anxiety (FASA) | Measured over the course of 6 months (14 months including follow-up)
  A parent-rated measure of parental accommodation to the child's anxiety
Trimbos/iMTA questionnaire for Costs associated with Psychiatric Illness (TiC-P) - Child version | Measured over the course of 6 months (14 months including follow-up)
  A parent-rated measure of direct and indirect costs related to psychiatric illness in children
The Negative Effects Questionnaire (NEQ) | Measured only at post-treatment
  A self-rated measure of treatment related adverse and unwanted events
Internet intervention Patient Adherence Scale (iiPAS) | Measured at mid-treatment (week 5) and at post-treatment (week 10)
  A clinician-rated measure of adherence to the allocated treatment
School absenteeism | Measured over the course of 6 months (14 months including follow-up)
  A parent-rated measure of the frequency of school absenteeism

CONTACTS AND LOCATIONS:
Overall Officials: Eva Serlachius, PhD, MD, Principal Investigator — Karolinska Institutet
Locations (1):
- BUP KFE, Stockholm, Stockholms County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nordh M, Wahlund T, Jolstedt M, Sahlin H, Bjureberg J, Ahlen J, Lalouni M, Salomonsson S, Vigerland S, Lavner M, Ost LG, Lenhard F, Hesser H, Mataix-Cols D, Hogstrom J, Serlachius E. Therapist-Guided Internet-Delivered Cognitive Behavioral Therapy vs Internet-Delivered Supportive Therapy for Children and Adolescents With Social Anxiety Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2021 Jul 1;78(7):705-713. doi: 10.1001/jamapsychiatry.2021.0469. PMID 33978699